CLINICAL TRIAL: NCT04587063
Title: Evaluation of an Email Intervention Promoting Enrollment in Mail-order Pharmacy
Brief Title: Evaluation of Emails Promoting Mail-order Pharmacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-0482
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Health Care Utilization
Keywords: Pharmacy; Postal Service; Electronic Mail; Communication; Economics, Behavioral; Psychology; Loss Frames; Fear Appeals
MeSH Terms: conditions — Patient Acceptance of Health Care; Communication; Behavior

STUDY DESIGN:
Intervention Model Description: 1 x 5 design
Who Masked: Participant, Care Provider
Masking Description: Participants and providers are not aware that different mailer versions exist, and they do not know what elements in the letter are being tested.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Standard Email (Active Comparator): The "standard of care" email is the same as one used in prior outreach efforts at the health system, emphasizing reduced cost for medications and convenience.
  Interventions: Behavioral: Highlighting Cost Savings and Convenience
- Email with Healthcare Cost Savings (Experimental): The email emphasizes future reductions in healthcare costs due to increased adherence with mail-order pharmacy, in addition to mentioning reduced prices for medications. It also uses fear appeals by stating the risk of hospital stays and how mail-order pharmacy could be an easily-achievable way to avoid this negative consequence.
  Interventions: Behavioral: Fear Appeals; Behavioral: Message about Future Healthcare Costs; Behavioral: Highlighting Cost Savings and Convenience
- Email with Endorsement (Experimental): The email is a letter from a doctor at the health system's health plan--who may been seen as a trusted source of information--encouraging the benefits of using a mail-order pharmacy.
  Interventions: Behavioral: Endorsement from a Doctor; Behavioral: Highlighting Cost Savings and Convenience
- Email with Comparison Table (Experimental): The email includes a table comparing the benefits and drawbacks of mail-order and chain pharmacies, which appeals to their sense of agency and allows them to make the choice that best suits them.
  Interventions: Behavioral: Comparison Table; Behavioral: Highlighting Cost Savings and Convenience
- No Contact (No Intervention): Members do not receive an email.

INTERVENTIONS:
Behavioral: Fear Appeals — Email
  Arms: Email with Healthcare Cost Savings
Behavioral: Message about Future Healthcare Costs — Email
  Arms: Email with Healthcare Cost Savings
Behavioral: Endorsement from a Doctor — Email
  Arms: Email with Endorsement
Behavioral: Comparison Table — Email
  Arms: Email with Comparison Table
Behavioral: Highlighting Cost Savings and Convenience — Email
  Arms: Email with Comparison Table; Email with Endorsement; Email with Healthcare Cost Savings; Standard Email

SUMMARY:
In this evaluation, four versions of emails will be sent to eligible health plan members who are not currently enrolled in the health system's mail-order pharmacy. A control group will not receive any communication. The researchers hypothesize that the use of content informed by behavioral nudge theory in the emails should lead to increased enrollment in the health system's mail-order pharmacy.

DETAILED DESCRIPTION:
The utilization of a mail-order pharmacy can increase adherence to medications. The health system's mail-order pharmacy (from here, simply referred to as mail-order pharmacy) can also provide reduced costs for medications. Ongoing outreach efforts involve sending emails and other communications encouraging enrollment in Geisinger's mail-order pharmacy to eligible members of the system's health plan (i.e., those who take maintenance medications). The study will compare a standard promotional email from these outreach efforts, as well as three new emails with content informed by behavioral science research, against a no-contact control arm and each other.

ELIGIBILITY:
Inclusion Criteria:

* An active member of the health plan (Medicare, Commercial, or Exchange)
* Currently prescribed maintenance medications
* Not currently subscribed to the health system's mail-order pharmacy
* Has an email on record

Exclusion Criteria:

* Explicitly opted out of receiving emails from the health system
* Only has eligible current prescriptions for fewer than 28 days
* Only has prescriptions that cannot be sent via mail-order pharmacy (e.g., antidepressants, specialty-tier drugs)
* Is a Medicare member in the coverage gap
* Shares an email address with another selected participant (who was randomly chosen for inclusion among all those sharing the same email address)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5266 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
Mail-order Pharmacy Enrollment | 1 week from the intervention
  Binary variable indicating if there was an enrollment in the health system's mail order pharmacy

SECONDARY OUTCOMES:
Email Opens | 1 week from the intervention
  Binary variable indicating if the email was opened
Email Link Click | 1 week from the intervention
  Binary variable indicating if the link to the mail-order pharmacy website was clicked
Email Unsubscribes | 1 week from the intervention
  Binary variable indicating if the recipient requested to unsubscribe from receiving emails from the health system

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings. The PI did not examine or analyze any data from this study prior to this registration.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.